CLINICAL TRIAL: NCT06311396
Title: Development of a Neuronal Microscope for Cell Characterization and Manipulation (Neuronal micRoscopy for cEll Behavioral Examination and mAnipuLation)
Brief Title: Development of a Neuronal Microscope
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Valenti:, Luca Vittorio Carlo Valenti, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REVEAL
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Models, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuronal micRoscopy for cEll behaVioural Examination and mAnipuLation (Experimental): validate the ability of a neuronal microscope to decipher the biomechanism at the origin of liver cancer, especially addressing the problem of biological heterogeneity
  Interventions: Genetic: genetic model

INTERVENTIONS:
Genetic: genetic model — Create a complete molecular-level description of the heterogeneous population of cells that are capable of giving rise to tumor transformation in the liver.

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common type of primary liver cancer and is a leading cause of cancer-related death worldwide. The prognosis of HCC remains poor, with a 5-year survival rate of 18%. Risk factors for HCC include viral infection, autoimmune hepatitis, chronic alcohol use or metabolic fatty liver disease, obesity, and diabetes mellitus.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common type of primary liver cancer and is a leading cause of cancer-related death worldwide. The prognosis of HCC remains poor, with a 5-year survival rate of 18%. Risk factors for HCC include viral infection, autoimmune hepatitis, chronic alcohol use or metabolic fatty liver disease, obesity, and diabetes mellitus. Furthermore, alterations and chronic inflammation of the microenvironment can facilitate the transformation of normal liver stem cells into precancerous tumor stem cells. All these underlying pathogenic stimuli can induce a spectrum of genetic and epigenetic modifications, which are involved in the cell cycle, cell growth and regulation of adhesion. Therefore, heterogeneity and tumor priming potential arise from a combination of both endogenous and exogenous factors. However, current in vitro models, based on conventional hepatoma and hepatocarcinoma cell lines, fail to recapitulate key characteristics of tumor tissue such as three-dimensional tissue architecture, cellular heterogeneity, and cell-cell interactions. Organoids, which are 3D cellular structures generated from induced pluripotent stem cells and adult tissue-resident stem cells, have recently been exploited to overcome the limitations of 2D cell culture systems, emerging as powerful tools for studying human diseases. Therefore, organoid structures stably preserve the genetic information of autologous tissue by mimicking the pathological state of the tissue itself.

ELIGIBILITY:
Inclusion Criteria:

Patients aged >18 years:

* undergoing surgical cholecystectomy, liver resection for hepatocellular carcinoma (both intra-tumoral and extra-tumoral tissues) or whole liver explants;
* who have given consent to participate in the study.

Exclusion Criteria:

• positivity for chronic viral hepatitis (HCV-RNA and HBsAg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Isolation of epithelial cells | January 2021 - January 2025
  Isolation of epithelial cells to ultimately generate models of major hepatocellular carcinoma cell populations in three-dimensional culture environment, called liver organoids, and molecular characterization of the generated models.
Omics studies and functional morphological studies | January 2021 - January 2025
  * Knowledge of the behavioral and morphological differences between physiological and tumor hepatocytes;
  * Knowledge of the molecular mechanisms underlying cellular level observations exploiting "omics" scale assessments and CRISPR-Cas9 genetic engineering

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT06311396/Prot_SAP_000.pdf